CLINICAL TRIAL: NCT04237974
Title: Evaluation of Different Prognostic Tools in Patients With Acute Pulmonary Thromboembolism
Brief Title: Prognostic Tools in Patients With Acute Pulmonary Thromboembolism.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amal Abdallah Abd Elrahman, assistant lecturer, Assiut University
Other Study IDs: pulmonary embolism prognosis
Record Dates: First submitted 2020-01-09; First posted 2020-01-23 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: computed tomography pulmonary angiography — The radiological severity of pulmonary embolism will be assessed by using the computed tomography pulmonary arterial obstruction index (CT-PAOI)
  Other Names: echocardiography

SUMMARY:
Acute pulmonary embolism (PE) is a serious disease associated with high mortality rates despite advanced therapeutic options. The treatment options depend on the severity of the disease and the short - term mortality varies widely from 2 to 95%, depending on the severity of the condition

DETAILED DESCRIPTION:
Acute pulmonary embolism (PE) is a serious disease associated with high mortality rates despite advanced therapeutic options. The treatment options depend on the severity of the disease and the short - term mortality varies widely from 2 to 95%, depending on the severity of the condition.

Initial risk stratification of patients with PE could be based on clinical indicators. The presence of shock and hypotension is the most important clinical sign of poor prognosis. Other clinical variables, associated with poor prognosis are age over 70 years, history of bed rest over five days, cancer, chronic obstructive pulmonary disease, renal failure, heart failure, and tachycardia .

Echocardiography represents the most useful imaging tool in everyday clinical practice to show right ventricular dysfunction (RVD) because of its noninvasive nature and relative low cost. RVD assessed on echocardiography has been described as one of the strongest predictor of early mortality in PE .

Currently, computed tomography pulmonary angiography (CTPA) represents the diagnostic gold standard for PE. Additionally, CTPA was used to evaluate the prognosis by determining the distribution and severity of vascular obstruction of clots in pulmonary circulation; this is called computed tomography pulmonary artery obstruction index (CT-PAOI). CTPA was also suggested as a predictor of RVD .

In addition to the clinical findings and the imaging abnormalities, there are several biomarkers and indicators that can be used to predict severity and prognosis in patients with PE. These biomarkers include troponin and brain natriuretic peptide (indicators of RVD and myocardial damage), D-dimer, C-reactive protein, arterial blood gases parameters and complete blood count (CBC) parameters. However, some of these biomarkers have not been widely studied and are not commonly used although they are readily available and cheaper for developing countries.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years) who will be diagnosed as acute pulmonary embolism based on computed tomography pulmonary angiography (CTPA) and not yet treated.

Exclusion Criteria:

1. Age less than 18 years.
2. Patients with known hematological disorders.
3. Patients with history of recent blood transfusion (within 3 weeks).
4. Patients receive anti-platelet and/or anticoagulant medications.
5. Patients receive immunosuppressive drugs.
6. Patients with known cardiopulmonary diseases other than the pulmonary embolism.
7. Patients with known active infectious diseases or immunological diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted at the Chest Department and Respiratory Intensive Care Unit (RICU) at Assiut University Hospital.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
prognostic importance of computed tomography pulmonary artery obstruction index (CT-PAOI) | 2 years
  To calculate the CT-PAOI, the arterial tree of each lung was considered to have 10 segmental arteries . The presence of an embolus in a segmental artery was scored 1 point. Central or paracentral emboli were scored a value equal to the number of segmental arteries arising distally. Depending on the degree of vascular obstruction a weighting factor was assigned to each value (0, no thrombus 1, partial occlusion and 2, total occlusion). Isolated subsegmental embolus was considered as a partially occluded segmental artery and was assigned a value of1. Thus, the PAOI could vary from 1 to 40 points per patient. Dividing the patient score by the maximal total score and multiplying the result by 100 calculated the percentage of vascular obstruction, Based on the which, patients were then divided into three groups (<15% versus 15-50% versus >50%).
prognostic importance of White blood cell count(WBC) . | 2 years
  * white blood cell count (number/cubic milliliter)
prognostic importance of polymorphonuclear cell count | 2 years
  -polymorphonuclear cell count (number/cubic milliliter)
prognostic importance of lymphocyte cell count | 2 years
  -lymphocyte cell count (number/cubic milliliter)
prognostic importance of a D-dimer level | 2 years
  - D-dimer level (microgram/liter)
prognostic importance of Troponin level | 2 years
  -Troponin level (nanogram/milliliter)
prognostic importance of C-reactive protein | 2 years
  - C-reactive protein (milligram /liter)
prognostic importance of arterial blood gases while the patients are breathing room air. | 2 years
  -Partial pressure of oxygen tension (millimeter mercury)
prognostic importance of hemoglobin level | 2 years
  -hemoglobin level (gram/deciliter)
prognostic importance of platelet cell count | 2 years
  -platelet cell count (number/cubic milliliter)
prognostic importance of red cell distribution width | 2 years
  -red cell distribution width (%)

CONTACTS AND LOCATIONS:
Overall Officials: Yousef A Yousef, Professor, Principal Investigator — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt

REFERENCES:
- [Background] Cohen AT, Agnelli G, Anderson FA, Arcelus JI, Bergqvist D, Brecht JG, Greer IA, Heit JA, Hutchinson JL, Kakkar AK, Mottier D, Oger E, Samama MM, Spannagl M; VTE Impact Assessment Group in Europe (VITAE). Venous thromboembolism (VTE) in Europe. The number of VTE events and associated morbidity and mortality. Thromb Haemost. 2007 Oct;98(4):756-64. doi: 10.1160/TH07-03-0212. PMID 17938798
- [Background] Goldhaber SZ, Visani L, De Rosa M. Acute pulmonary embolism: clinical outcomes in the International Cooperative Pulmonary Embolism Registry (ICOPER). Lancet. 1999 Apr 24;353(9162):1386-9. doi: 10.1016/s0140-6736(98)07534-5. PMID 10227218
- [Background] Becattini C, Agnelli G. Acute pulmonary embolism: risk stratification in the emergency department. Intern Emerg Med. 2007 Jun;2(2):119-29. doi: 10.1007/s11739-007-0033-y. Epub 2007 Jul 9. PMID 17619833
- [Background] Goldhaber SZ. Echocardiography in the management of pulmonary embolism. Ann Intern Med. 2002 May 7;136(9):691-700. doi: 10.7326/0003-4819-136-9-200205070-00012. PMID 11992305
- [Background] Qanadli SD, El Hajjam M, Vieillard-Baron A, Joseph T, Mesurolle B, Oliva VL, Barre O, Bruckert F, Dubourg O, Lacombe P. New CT index to quantify arterial obstruction in pulmonary embolism: comparison with angiographic index and echocardiography. AJR Am J Roentgenol. 2001 Jun;176(6):1415-20. doi: 10.2214/ajr.176.6.1761415. PMID 11373204
- [Background] Lega JC, Lacasse Y, Lakhal L, Provencher S. Natriuretic peptides and troponins in pulmonary embolism: a meta-analysis. Thorax. 2009 Oct;64(10):869-75. doi: 10.1136/thx.2008.110965. Epub 2009 Jun 11. PMID 19525265
- [Background] Becattini C, Lignani A, Masotti L, Forte MB, Agnelli G. D-dimer for risk stratification in patients with acute pulmonary embolism. J Thromb Thrombolysis. 2012 Jan;33(1):48-57. doi: 10.1007/s11239-011-0648-8. PMID 22109384
- [Background] Abul Y, Karakurt S, Ozben B, Toprak A, Celikel T. C-reactive protein in acute pulmonary embolism. J Investig Med. 2011 Jan;59(1):8-14. doi: 10.2310/jim.0b013e31820017f2. PMID 21218608
- [Background] Subramanian M, Ramadurai S, Arthur P, Gopalan S. Hypoxia as an independent predictor of adverse outcomes in pulmonary embolism. Asian Cardiovasc Thorac Ann. 2018 Jan;26(1):38-43. doi: 10.1177/0218492317746252. Epub 2017 Dec 20. PMID 29260572